CLINICAL TRIAL: NCT04419662
Title: Evaluation of Patients After Cardiac Surgery: Novel Ultrasound Parameters for Quantification of Renal Perfusion & Analysis of Phenylephrines' Effect on Invasive Haemodynamics and Echocardiographic Measures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Johan Fridolf Hermansen, Principal Investigator, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-10-72-40-20; 2020-000573-25 (EudraCT Number)
Record Dates: First submitted 2020-04-30; First posted 2020-06-05 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Ultrasonography, Renal; Cardiac Surgery; Hemodynamics; Phenylephrine; Renal Perfusion; Echocardiography; Anesthesia
MeSH Terms: interventions — Phenylephrine; Patient Positioning

STUDY DESIGN:
Masking Description: Ultrasound analysis is performed offline and details on participants and time of measurement are blinded for the person doing the analysis. The personnel responsible for obtaining data will not be blinded towards any of the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients included (Experimental)
  Interventions: Drug: Phenylephrine; Other: Combination of PEEP and positioning

INTERVENTIONS:
Drug: Phenylephrine — Three time points: before, during and 20-30 minutes after infusion of phenylephrine.
  Patients will receive an infusion of up to 1 mcg/kg/min phenylephrine intravenously to raise mean arterial pressure with 20 mmHg for 10 minutes. Infusion of phenylephrine will start at 0.1 mcg/kg/min with subsequent titration to effect.
Other: Combination of PEEP and positioning — Six time points based on combinations of the following:
  Three different levels of PEEP (as set on the ventilator): 0, 6 and 12 mmHg. Two different positions: 1) torso elevated 30 degrees, legs horizontal and 2) torso horizontal, legs elevated 30 degrees.

SUMMARY:
To investigate the influence of PEEP (Positive end-expiratory pressure), changes in preload (patient position) and changes in afterload (phenylephrine) on ultrasound measures of renal perfusion in patients after uncomplicated cardiac surgery.

To investigate the effects of phenylephrine on both invasive measures of the systemic- and pulmonary circulation and, secondarily, to assess the induced changes in echocardiographic indices of left- and right ventricular systolic- and diastolic function.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥ 18 years scheduled for open elective cardiac surgery at the Department of Cardiothoracic & Vascular Surgery, Aarhus University Hospital.

Exclusion Criteria:

* Insufficient ultrasonographic imaging of the kidneys
* Known morphological kidney disease
* Preoperative dialysis
* Chronic atrial fibrillation
* Planned mitral valve surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Renal arterial resistive index (RI). | 75 minutes
The ratio SVR/PVR (systemic vascular resistance/pulmonary vascular resistance) | 75 minutes

SECONDARY OUTCOMES:
Renal venous impedance index. | 75 minutes
Renal venous stasis index. | 75 minutes
Portal vein pulsatility fraction. | 75 minutes
Cardiac output | 75 minutes
Arterial blood pressure, central venous pressure, pulmonary blood pressure, pulmonary capillary wedge pressure. | 75 minutes
Transoesophageal measurement of left and right ventricular function 1 | 75 minutes
  Systolic measure (ejection fraction (EF))
Transoesophageal measurement of left and right ventricular function 2 | 75 minutes
  Systolic measure (s')
Transoesophageal measurement of left and right ventricular function 3 | 75 minutes
  Systolic measure (strain)
Transoesophageal measurement of left and right ventricular function 4 | 75 minutes
  Diastolic measures (E, A,)
Transoesophageal measurement of left and right ventricular function 5 | 75 minutes
  Diastolic measures (e', a')
Transoesophageal measurement of left and right ventricular function 6 | 75 minutes
  Diastolic measure (deceleration time)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Juhl-Olsen, MD, PhD, Study Chair — Aarhus University Hospital; Johan F Hermansen, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Department of Anaesthesiology, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Juhl-Olsen P, Berg-Hansen K, Norskov J, Enevoldsen J, Hermansen JL. The haemodynamic effects of phenylephrine after cardiac surgery. Acta Anaesthesiol Scand. 2023 Aug;67(7):869-876. doi: 10.1111/aas.14256. Epub 2023 Apr 25. PMID 37186094
- [Derived] Hermansen JL, Norskov J, Juhl-Olsen P. Effects of changes in position, positive end-expiratory pressure and mean arterial pressure on renal, portal and hepatic Doppler ultrasound perfusion indices: a randomized crossover study in cardiac surgery patients. J Clin Monit Comput. 2022 Dec;36(6):1841-1850. doi: 10.1007/s10877-022-00834-0. Epub 2022 Mar 1. PMID 35230558